CLINICAL TRIAL: NCT05698745
Title: Prospective Study of the Natural History, Immunological and Genetic Characteristics of Preclinical Inflammatory Bowel Disease
Brief Title: Immunological Characteristics of Preclinical IBD
Status: Recruiting | Type: Observational
Sponsor: Grupo Espanol de Trabajo en Enfermedad de Crohn y Colitis Ulcerosa (Other)
Responsible Party: Sponsor
Other Study IDs: EARLY
Record Dates: First submitted 2023-01-10; First posted 2023-01-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Crohn Disease; Ulcerative Colitis; IBD
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, serum, plasma, urine, stools, small/large bowel tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A (preclinical IBD): asymptomatic patients with a new diagnosis of IBD during the colorectal cancer screening programme meeting all inclusion and none of the exclusion criteria (n=350).
  Interventions: Procedure: bioespecimen samples
- Cohort B (control): new-onset symptomatic IBD (n=80) - patients with a symptomatic debut of IBD in the last 3 months, naïve to immunosuppressants and biologic agents.
  Interventions: Procedure: bioespecimen samples
- Cohort C (control): healthy controls (n=20): patients with a normal screening colonoscopy, with no signs of IBD after a detailed evaluation of the ileum and colon, will be included.
  Interventions: Procedure: bioespecimen samples

INTERVENTIONS:
Procedure: bioespecimen samples — Blood, serum, plasma, urine, stools, small/large bowel tissue.

SUMMARY:
The purpose of this study is to evaluate disease progression, in terms of development of symptomatic disease and complications associated with IBD (e.g. fistula, abscess, stricture).

DETAILED DESCRIPTION:
This is a prospective, observational, multicenter, collaborative research project that will explore the earlier stages of IBD, before the onset of the first symptoms of the disease. This novel approach constitutes an innovative strategy on the research on the natural history of the disease. The study will be carried out based on colorectal cancer screening colonoscopies, recruiting all patients with a new diagnosis of IBD in this setting. These patients will undergo follow-up visits every 6 months for 10 years and the clinical information will be enriched with longitudinal multi-omic analyses.

Two additional control groups will be identified, including patients with new-onset symptomatic IBD in the last 3 months and healthy controls (with normal screening colonoscopy).

ELIGIBILITY:
Inclusion criteria

Patients from cohort A will be included if they fulfill all the following inclusion criteria:

* Male or female ≥18 years of age at baseline.
* New diagnosis of IBD during a CRC screening colonoscopy, based on the criteria from the European Crohn's and Colitis Organization (33, 34).
* Presence of a chronic inflammatory infiltrate and histological diagnosis compatible with IBD.
* The patient must be asymptomatic at diagnosis and without previous symptoms suggestive of IBD.
* Time interval between the index colonoscopy and the baseline visit up to 3 months.

Patients from cohort B will be included if they fulfill all the following inclusion criteria:

* Male or female ≥18 years of age at baseline.
* Recent diagnosis of IBD, with <3 months from symptoms onset.
* Time interval between the index colonoscopy and the baseline visit up to 3 months.

Patients from cohort C will be included if they fulfill all the following inclusion criteria:

* Male or female ≥18 years of age at baseline.
* No endoscopic signs of IBD after a complete ileo-colonoscopy within the CRC screening program.
* Time interval between the index colonoscopy and the baseline visit up to 3 months.

Exclusion criteria

Patients from cohort A will be excluded if they fulfill any the following exclusion criteria:

* Identification of any enteropathogen in the stool culture.
* Isolated findings of acute inflammatory infiltrate without signs of chronicity.
* Previous or current diagnosis of microscopic colitis.
* Alteration in biomarkers in blood or stool will not constitute an exclusion criterion.

Patients from cohort B will be excluded if they fulfill any the following exclusion criteria:

- Previous use of immunomodulators or biologics for any condition.

Patients from cohort C will be excluded if they fulfill any the following exclusion criteria:

* Any gastrointestinal symptoms at baseline.
* Previous use of immunomodulators or biologics for any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with a new diagnosis of IBD
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2038-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease progression | 10 years
  Development and type of new-onset symptoms during follow-up (mainly diarrhea, abdominal pain, and rectal bleeding).
Disease progression | 10 years
  Time to development of symptomatic disease during follow-up.
- IBD characteristics | 10 years
  * Type (CD or UC)
  * Disease extent (CD or UC) according to Montreal classification
  * CD phenotype at diagnosis (Montreal classification)
  * Endoscopic characteristics at diagnosis (both CD and UC): type of lesions, distribution, and extent
  * Presence and type (simple, complex fistula or abscess) of perianal disease at diagnosis and during follow-up
Omic findings | 10 years
  proteomic, transcriptomic, serologic, microbiota, and tissue data

SECONDARY OUTCOMES:
IBD characteristics: | 10 years
  * Development and time to development of changes in CD disease location, according to Montreal classification.
  * Development and time to development of new-onset or stricturing, penetrating or perianal complications, defined as changes in CD phenotype (Montreal classification)
  * Development of proximal disease extension in UC
  * Laboratory parameters: FOBT levels at diagnosis, and CRP, hemoglobin, albumin, fecal calprotectin at diagnosis and during follow-up.
Changes in endoscopic features during follow-up | 10 years
Microscopic characteristics at diagnosis | 10 years
Clinical disease activity during follow-up | 10years
Development and time to development of need for medical or surgical therapy during follow-up | 10years
Development and time to development of extraintestinal manifestations during follow-up | 10years
Type of extraintestinal manifestations during follow-up | 10years

CONTACTS AND LOCATIONS:
Overall Officials: Iago Rodriguez Lago, MD, Principal Investigator — Spanish Working Group on Crohn's disease and ulcerative colitis (GETECCU)
Locations (24):
- Spain (24):
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela, A Coruña
  - Hospital General Universitario Dr. Balmis, Alicante, Alicante
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Sant Joan Despí Moisès Broggi, Barcelona, Barcelona
  - Althaia, Xarxa Assistencial Universitària de Manresa, Manresa, Barcelona
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Basurto, Bilbao, Bilbao
  - Hospital Universitario de Burgos, Burgos, Burgos
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Complejo Hospitalario Universitario de Ourense, Ourense, Ourense
  - Hospital Álvaro Cunqueiro (Complejo Hospitalario Universitario de Vigo), Vigo, Pontevedra
  - Hospital Universitario de Cabueñes, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Hospital Universitario Clínico de Valencia, Valencia, Valencia
  - Hospital Univeristario y Politécnico La Fe, Valencia, Valencia
  - Hospital Universitario Río Hortega, Valladolid, Valladolid
  - Hospital Universitario de Galdakao, Galdakao, Vizcaya
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rodriguez-Lago I, Marigorta UM, Mateos B, Manosa M, Marquez-Mosquera L, Menchen L, Rodriguez-Moranta F, Alonso I, Aguas M, Alonso-Galan H, Borras P, Castro B, Domenech E, Ferreiro-Iglesias R, de Francisco R, Garcia-Alonso FJ, Garcia N, Garcia-Bosch O, Gargallo C, Gisbert JP, Iglesias E, Mesonero F, Ortiz de Zarate J, Ramos L, Sainz E, Ladron P, Suria C, Ferrer CS, Tejido C, Varela P, Vicente R, Zabana Y, Castany G, Rodriguez E, Gutierrez A, Barreiro-de Acosta M. Natural history, immunological and genetic characteristics of preclinical inflammatory bowel disease (EARLY): study protocol for a prospective cohort study. Therap Adv Gastroenterol. 2025 May 12;18:17562848251338647. doi: 10.1177/17562848251338647. eCollection 2025. PMID 40365077